CLINICAL TRIAL: NCT05770440
Title: Impact of COVID-19 on Lung Function in COPD Patients
Acronym: EspirCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Other Study IDs: 243
Record Dates: First submitted 2023-03-14; First posted 2023-03-15 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: COPD; COVID-19
Keywords: COPD; COVID-19; Lung Function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patient with COPD and at least 1 SARS-Cov2 Infection
- Group 2: Patient with COPD and no SARS-COV2 Infection

SUMMARY:
Background: In 2019, a novel coronavirus (SARS-COV2) was detected in Wuhan, China as a cause of acute respiratory distress syndrome (COVID-19). Other previous coronaviruses (SARS and MERS) have caused respiratory sequelae (pulmonary fibrosis) demonstrable by tomography and lung function tests. These alterations have begun to be detected in patients who have survived COVID-19.

Hypotheses: SARS-COV2 infection accelerates the deterioration of lung function in patients with Chronic Obstructive Pulmonary Disease (COPD).

Objectives: To analyze the evolution of lung function in COPD patients diagnosed with COVID-19, while comparing it with COPD patients without COVID-19 disease.

Methodology: Cohort study. The COPD-COVID-19 cohort will consist of the COPD population with and without COVID-19. Previous pulmonary function data will be collected and 2 prospective visits (baseline and follow-up) with clinical assessments and functional tests will be performed. In the event that the participant suffers from COVID-19 during the follow-up, an additional visit will be performed 3 months after the diagnosis, and the final visit will take place 12 months after this additional visit.

Determinations: Study factor: diagnosis of COVID-19. Response variable: change in the forced expiratory volume in the first second (FEV1) measured at the start of the study and after 1 year of this first assessment, considering also the basal FEV1 (before March 2020). Other variables: socio-demographic, clinical, functional and treatment.

Expected results: Greater decrease in FEV1 in COPD patients with COVID-19, Applicability and Relevance: The proactive detection of functional sequelae will allow early treatment, including pulmonary rehabilitation, with the aim of improving the quality of life of these patients.

DETAILED DESCRIPTION:
BACKGROUND Million people have suffered COVID-19 in Spain, being the respiratory system the most affected in many patients. Some studies, with short follow-up periods, have reported an impairment of respiratory function after pneumonia due to COVID-19.

COPD patients are considered a risk group for SARS-CoV-2 infection and poor prognosis in case of COVID-19; furthermore, in them respiratory function is usually already impaired.

It is in this context that a study of the evolution of the lung function of COPD patients who have overcome COVID-19 is proposed. It is hypothesized that COVID-19 accelerates the deterioration of lung function in patients with COPD.

AIMS

General:

To analyze the evolution of lung function in COPD patients who have suffered mild or moderate COVID-19, while comparing it with that of patients with COPD who have not.

Specific:

To analyze the influence of different variables, including the history of COVID-19, on the evolution of lung function in COPD patients.

METHODS

Design:

Cohort study in patients diagnosed with COPD. Two subgroups of participants will be distinguished:

1. COVID-19 group: Patients with COPD diagnosed with COVID-19 before recruitment or during the study period.
2. Non-COVID-19 group: Patients with COPD who have not suffered from COVID-19 either before or during the study

Sample size calculation:

To calculate the sample size, the dependent variable is considered the difference between basal FEV1 (corresponding to the last spirometry recorded in the clinical history, previous to the study start), FEV1 obtained at the first assessment, and final FEV1 (obtained at the second assessment, after one year).

Accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a bilateral contrast, 22 subjects in the first group and 88 in the second group are needed to detect a difference equal to or greater than 30 units (assuming a common SD of 59 [Vetsbo et al, 2021], a between-groups ratio of 1:4, a correlation between the first and second measurements of 0.75, and a loss-to-follow-up rate of 10%).

Recruitment of participants and inclusion procedure An information session will be held at the Primary Care Centres (PCC) in the territory to advise about the study, its characteristics and objectives. At least the person in charge of spirometry's performing will be offered to participate as a reference research person (RRP) of the study at that PCC.

Participants will be selected by consecutive sampling, by their reference professional (doctor or nurse), from the study start until the expected sample size is reached. According to guidelines recommendation, follow-up spirometry will be offered to all COPD patients who consult their primary care team, regardless of the reason for the consultation and as long as they have no contraindications for the test. In the same consultation, they will be offered participation in the study, they will be informed of the procedures and reasons for the study, and they will be given the information sheet and informed consent sheet. If they decide to sign consent, they will be recruited by the RRP when they come to perform forced spirometry.

RRP will then check if participants have been diagnosed of COVID-19 through any registered test (PCR, ART and/or serology) with a positive result, and will record this information in the ad hoc data collection book (DCB), along with socio-demographic variables. Spirometry will be performed to participants without a history of COVID-19, and to those with a diagnosis of COVID-19 registered more than 3 months ago; spiromètric parameters (FEV1, FVC...) will be recorded at DCB. In participants with COVID-19 diagnosis in the previous three months, spirometry and initial evaluation will be scheduled after 3 months of diagnosis, according to the local protocol.

First assessment In the first assessment, data will be collected from electronic medical records (comorbidities, medications); moreover, physical examination and clinical assessment tests will be undertaken. In PCC that have adequate facilities, the 6-minute walk test (6MWT) will be carried out. This test is included in the monitoring of the COPD patient, as part of the BODE index, with implications on the severity and prognosis of the disease. If the 6MWT cannot be performed, as an alternative to the BODE index, the BODEx index (which replaces the 6MWT for the number of COPD exacerbations in the previous 12 months) will be calculated.

Finally, RRP will give an appointment to the participants for the final evaluation, one year later, unless they are diagnosed with COVID-19 in that period; in that case, participants will contact with RRP for new assessment three months after COVID-19 diagnosis, and will change from the non-COVID-19 cohort subgroup to the COVID-19 cohort subgroup Follow-up After the first spirometry and first assessment, all participants will have a second follow-up visit. In patients who do not suffer from COVID-19 during the follow-up period, this final visit will take place 12 months after the inclusion in the study. In patients who present COVID-19 during follow-up, this second assessment will be taken out 15 months after the diagnosis of COVID-19. The content of this follow-up visit will be the same as that of the first assessment, including records of spirometric parameters, that will allow to analyse outcome measures.

Statistical analysis A first descriptive data analysis shall be carried out, providing absolute and relative frequencies for categorical variables, and mean, and standard deviation (or median, and interquartile range, in case they are not distributed according to normal distribution) for continuous variables.

Differences in successive measurements of FEV1 (baseline, initial and final) between the subgroups with and without COVID-19 shall be compared using the ANOVA test for paired samples, or the Kruskal-Wallis test if the FEV1 values are not distributed according to normal law.

The influence of other variables of interest on the evolution of the FEV1 value will be analyzed by means of mixed linear models, considering as fixed factors: background of COVID-19 (yes/no), all those that have shown significant differences in the bivariate analysis (possible confounding variables), and those recognized as clinically relevant; and as random factors: patients and patient visits.

Study difficulties and limitations Due to the type of sampling, it cannot be guaranteed that COPD patients without COVID-19 are similar to COPD with COVID-19; in any case, we will report the comparative analysis of the study variables between the two cohort subgroups.

As an observational study, the estimation of the contribution of the study variables to a greater deterioration of lung function may be influenced by confounding variables that have not been considered, and therefore not be rigorous.

Lastly, due to change of diagnostic protocol COVID-19 from March 2022 (the screening was stopped in asymptomatic and in symptomatic but not vulnerable people, including COPD persons), It could be that some members of the non-COVID-19 group have passed a mild, undiagnosed COVID-19.

Expected results and relevance If a greater decrease in respiratory function is observed in COPD patients who have suffered from COVID-19, close monitoring, and early preventive and treatment measures could be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* - Patients over 18 years of age with a diagnosis of COPD (register code J44.9 according to the 10th edition of the International Classification of Diseases, ICD-10).
* Fulfilling spirometric diagnostic criteria prior to January 1, 2020.
* Last valid spirometry after January 1, 2017.
* Availability and acceptance of the follow-up proposed in the study.

Exclusion Criteria:

* - Lack of basal spirometry recorded in the Computerized Primary Care Clinical History (eCAP).
* Spirometry results not compatible with COPD.
* Having suffered severe and/or critical COVID: It will be considered in accordance with the NICE classification:
* (1) Serious illness: Patients with clinical signs of pneumonia (fever, cough, dyspnea, rapid breathing) plus one of the following seriousness: a) respiratory frequency greater than 30 breaths per minute; b) severe respiratory distress or; c) SatO2 lower than 90% in ambient air.
* (2) Critical illness: Includes patients with Acute Respiratory Distress Syndrome (ARDS) and/or patients with septic shock and/or multi-organ disease.
* Any chronic or terminal condition that may make it difficult to carry out the necessary tests during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scope and period of study:
  Field of study: Primary Care; 20 primary care centers managed by the Catalan Health Institute in Camp de Tarragona.
  Study period: September 2022 to December 2024.
  Participants:
  Patients diagnosed with COPD, by means of spirometry (FEV1/FVC quotient <0.7 post-bronchodilation) before January 1, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in the first second (FEV1) | Baseline and 12 months
  This parameter shall be determined by spirometry after bronchodilator administration, and shall allow measurement of the degree of airway obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Albert Del Pozo-Niubó, MD, Principal Investigator — Institut Català de la Salut
Locations (1):
- Primary HealthCare Center of Falset, Falset, Tarragona, Spain

REFERENCES:
- [Background] Cherrez-Ojeda I, Gochicoa-Rangel L, Salles-Rojas A, Mautong H. [Follow-up of patients after COVID-19 pneumonia. Pulmonary sequelae]. Rev Alerg Mex. 2020 Oct-Dec;67(4):350-369. doi: 10.29262/ram.v67i4.847. Spanish. PMID 33631903
- [Background] Tabernero Huguet E, Urrutia Gajarte A, Ruiz Iturriaga LA, Serrano Fernandez L, Marina Malanda N, Iriberri Pascual M, Zalacain Jorge R. [Pulmonary Function in Early Follow-up of patients with COVID-19 Pneumonia]. Arch Bronconeumol. 2021 Jan;57:75-76. doi: 10.1016/j.arbres.2020.07.017. Epub 2020 Aug 1. No abstract available. Spanish. PMID 34629672
- [Background] Halpin DMG, Criner GJ, Papi A, Singh D, Anzueto A, Martinez FJ, Agusti AA, Vogelmeier CF. Global Initiative for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease. The 2020 GOLD Science Committee Report on COVID-19 and Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2021 Jan 1;203(1):24-36. doi: 10.1164/rccm.202009-3533SO. PMID 33146552
- [Background] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Background] Huang L, Yao Q, Gu X, Wang Q, Ren L, Wang Y, Hu P, Guo L, Liu M, Xu J, Zhang X, Qu Y, Fan Y, Li X, Li C, Yu T, Xia J, Wei M, Chen L, Li Y, Xiao F, Liu D, Wang J, Wang X, Cao B. 1-year outcomes in hospital survivors with COVID-19: a longitudinal cohort study. Lancet. 2021 Aug 28;398(10302):747-758. doi: 10.1016/S0140-6736(21)01755-4. PMID 34454673
- [Background] Leung JM, Niikura M, Yang CWT, Sin DD. COVID-19 and COPD. Eur Respir J. 2020 Aug 13;56(2):2002108. doi: 10.1183/13993003.02108-2020. Print 2020 Aug. PMID 32817205
- [Background] Maniscalco M, Ambrosino P, Fuschillo S, Stufano S, Sanduzzi A, Matera MG, Cazzola M. Bronchodilator reversibility testing in post-COVID-19 patients undergoing pulmonary rehabilitation. Respir Med. 2021 Jun;182:106401. doi: 10.1016/j.rmed.2021.106401. Epub 2021 Apr 13. PMID 33873099
- [Background] Salem AM, Al Khathlan N, Alharbi AF, Alghamdi T, AlDuilej S, Alghamdi M, Alfudhaili M, Alsunni A, Yar T, Latif R, Rafique N, Al Asoom L, Sabit H. The Long-Term Impact of COVID-19 Pneumonia on the Pulmonary Function of Survivors. Int J Gen Med. 2021 Jul 9;14:3271-3280. doi: 10.2147/IJGM.S319436. eCollection 2021. PMID 34267545
- [Background] Sanchez-Salcedo P, de Torres JP. BODE Index: A Good Quality of Life Marker in Chronic Obstructive Pulmonary Disease Patients. Arch Bronconeumol. 2015 Jul;51(7):311-2. doi: 10.1016/j.arbres.2015.03.003. Epub 2015 Apr 21. No abstract available. English, Spanish. PMID 25910549
- [Background] Soler-Cataluna JJ, Martinez-Garcia MA, Sanchez LS, Tordera MP, Sanchez PR. Severe exacerbations and BODE index: two independent risk factors for death in male COPD patients. Respir Med. 2009 May;103(5):692-9. doi: 10.1016/j.rmed.2008.12.005. Epub 2009 Jan 7. PMID 19131231
- [Background] Torres-Castro R, Vasconcello-Castillo L, Alsina-Restoy X, Solis-Navarro L, Burgos F, Puppo H, Vilaro J. Respiratory function in patients post-infection by COVID-19: a systematic review and meta-analysis. Pulmonology. 2021 Jul-Aug;27(4):328-337. doi: 10.1016/j.pulmoe.2020.10.013. Epub 2020 Nov 25. PMID 33262076
- [Background] Kerti M, Balogh Z, Kelemen K, Varga JT. The relationship between exercise capacity and different functional markers in pulmonary rehabilitation for COPD. Int J Chron Obstruct Pulmon Dis. 2018 Feb 28;13:717-724. doi: 10.2147/COPD.S153525. eCollection 2018. PMID 29535512
- [Background] Zhao YM, Shang YM, Song WB, Li QQ, Xie H, Xu QF, Jia JL, Li LM, Mao HL, Zhou XM, Luo H, Gao YF, Xu AG. Follow-up study of the pulmonary function and related physiological characteristics of COVID-19 survivors three months after recovery. EClinicalMedicine. 2020 Aug;25:100463. doi: 10.1016/j.eclinm.2020.100463. Epub 2020 Jul 15. PMID 32838236
- See also: Malaltia pulmonar Obstructiva crònica: guies de pràctica clínica. Barcelona: Institut Català de la Salut. — http://scientiasalut.gencat.cat/bitstream/handle/11351/4517/malaltia_pulmonar_obstructiva_cronica_guies_practica_clinica_2010_versio_breu.pdf?sequence=2&isAllowed=y
- See also: Recomanacions per a la realització d'espirometries a l'atenció primària en l'entorn COVID-19. Barcelona: Departament de Salut — https://scientiasalut.gencat.cat/handle/11351/6238
- See also: Global iniciative for Chronic Obstructive Lung Disease (GOLD). Pocket guide to COPD diagnosis, management, and prevention (2021 report) — http://goldcopd.org/wp-content/uploads/2020/11/GOLD-2021-POCKET-GUIDE-v1.0-16Nov20_WMV.pdf
- See also: Protocolo COVID ministerio Sanidad y Consumo España — http://www.mscbs.gob.es/profesionales/saludPublica/ccayes/alertasActual/nCov/documentos/Actualizacion_462_COVID-19.pdf
- See also: Clínica COVID Ministerio Sanidad y Consumo España — http://www.mscbs.gob.es/profesionales/saludPublica/ccayes/alertasActual/nCov/documentos/20210528_CLINICA.pdf